CLINICAL TRIAL: NCT07246915
Title: A Non-interventional, Extension Study on the Long-term Maintenance of Safety and Performance of the REVISYON SDS 100 Medical Device in Subjects With Mild-to-moderate Cataract
Brief Title: Long-term Safety & Performance of REVISYON SDS100 in Mild to Moderate Cataract: Extension Study (EB-CE-02)
Acronym: EB-CE-02
Status: Enrolling by invitation | Type: Observational
Sponsor: Edinburgh Biosciences Ltd (Industry)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Other Study IDs: EB-CE-02; QM75-OSP-001 (Other: Edinburgh Biosciences Ltd)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Age-related Cataract; Vision Loss; Cataract; Mild Cataract; Moderate Cataract
Keywords: REVISYON SDS 100; Visual acuity; EB-CE-02; EB-CE-01; Long-term safety; Non-interventional; Extension study; Cataract; Vision loss; LEDINBIO CE Device; Age-related Cataract
MeSH Terms: conditions — Vision Disorders; Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: The study population will consist of adult subjects with vision loss due to mild or moderate cataract, who were previously treated with the medical device in the EB-CE-01 study (one eye only, recorded as the study eye).
  The exclusion criteria are intended to protect subject safety and to ensure the integrity and validity of the clinical investigation by excluding subjects for whom participation may present undue risk.

SUMMARY:
A non-interventional, extension study on the long-term maintenance of safety and performance of the REVISYON SDS 100 medical device in subjects with mild-to-moderate cataract.

DETAILED DESCRIPTION:
This study is an ancillary study to the EB-CE-01 clinical investigation. No treatment or any study-specific intervention is foreseen for the study subcohort. This study is designed to evaluate the maintenance of safety and efficacy an average 20 months following the end of treatment of mild-to-moderate senile cataract with the medical device in the EB-CE-01 clinical investigation in the Romanian subcohort of subjects. Due to the long enrolment gap and different treatment intervals, the tracking of subjects provided a significant difference in the intervals since treatment completion among subjects.

Therefore, the study approach involves a single additional visit for subjects who initiated treatment, during which supplementary data will be collected from standard-of-care ophthalmological assessments.

In the initial EB-CE-01 study, treatment with the non-invasive medical device REVISYON SDS 100 was administered between April 2023 and December 2024 to 92 patients, all of whom were included in both the Full Analysis Set and the Safety Set. Best corrected visual acuity (BCVA) was assessed at 7 (±1) days, 28 (±4) days, and 84 (±10) days following the final treatment session (known as Visit 9). Treatment efficacy was evaluated at 7 (±1) days only, corresponding to one-week post-treatment.

In this extension study, prospective data will be collected to assess the incidence of any safety events and to evaluate the maintenance of best-corrected visual acuity (BCVA), cataract severity grade, and visual functioning at an additional follow-up visit. The following timepoints from the parent study will be used as reference: EB-CE-01 V0 (pre-treatment), EB-CE-01 V1-V9 (treatment visits), and EB-CE-01 V12 (last efficacy visit), which will serve as the baseline for the current extension study.

The main objective of the study is capturing any new clinically significant findings that meet the definition of an AE in accordance with EU MDR 2017/745 and ISO 14155:2020, as to generate robust safety findings in the pre-market stage.

As secondary objectives, the study will assess the mean change in best-corrected visual acuity (BCVA), the preservation of cataract severity grade, and the subjective evaluation of visual function using The Visual Function Index-14 (VF-14) relative to the last post-treatment assessment, defined at Visit 12 of the EB-CE-01 clinical investigation.

Study participants will be required to provide additional answers related to the visual functioning (VF-14 questionnaire), which will be administered in Romanian using linguistically validated versions. VF-14 questionnaire is a validated, brief questionnaire, including self-reported measures, designed to be completed within a few minutes, and is therefore not expected to constitute a burden or interfere with routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have initiated the EB-CE-01 study treatment phase in Romania
* Availability of complete retrospective data from the EB-CE-01 study- specifically from visit 12 assessment- including binocular BCVA, binocular LOCS III assessments, binocular slit-lamp assessment, and baseline assignment of the study eye.
* Be able and willing to follow instructions
* Subject whom the medical health history has been reviewed by the Investigator and medical records do not contraindicate the participation to the study. Note: Subjects who underwent cataract surgery in either eye will be allowed to participate

Exclusion Criteria:

* Subject unable to give voluntary written informed consent, is unlikely to cooperate or is legally incompetent, including subjects who are institutionalised by court or official order, or in a dependency relationship with sponsor, testing centre or investigator.
* Subject involved in other clinical investigation that may compromise the results of the study.
* Subjects developing mental illnesses that can influence their participation in the study (cognitive impairment, psychiatric condition, or neurological disorder).
* Any health condition which could interfere with the subject's ability to comply with the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult subjects, affected by vision loss due to early-stage cataract who had been assessed for BCVA and LOCS III nuclear grade and underwent treatment during the EB-CE-01 clinical investigation
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
A summary of adverse events | An average 20 months (following the end of treatment with the medical device initiated in the EB-CE-01 clinical investigation),
  A summary of adverse events collected over an average of 20 months following the end of treatment with the medical device initiated in the EB-CE-01 clinical investigation.
  The types of adverse events to be collected (AEs, SADEs, USADEs, AESIs, and SAEs) will be classified by type, severity, outcome, seriousness and causality).

SECONDARY OUTCOMES:
The mean change from Baseline post-treatment in Best Corrected Visual Acuity (BCVA), assessed using LogMAR scale | An average 20 months (following the end of treatment with the medical device initiated in the EB-CE-01 clinical investigation),
  Change in LogMAR = LogMAR (extended visit) - LogMAR (Visit 12, EB-CE-01 study)
Preservation of the cataract severity grade, assessed using LOCS III grading scale for nuclear domain beyond 3 months | An average 20 months (following the end of treatment with the medical device initiated in the EB-CE-01 clinical investigation),
  Change in LOCS III = LOCS III (extended visit) - LOCS III (Visit 12, EB-CE-01 study)
Subjective assessment of Visual function and Quality-of-life will be defined by the Visual Function Index-14 (VF-14) questionnaire data collected an average 20 months following the end of treatment with the medical device initiated in the EB-CE-01 study | An average 20 months (following the end of treatment with the medical device initiated in the EB-CE-01 clinical investigation),
  Change in Visual Function Index-14 (VF-14) Total Score (range 0-100, with higher scores representing better visual function) and changes in each of the 14 item-level scores (each item scored 0-4, with higher scores indicating less difficulty) from Visit 12 (EB-CE-01 study) to the extended follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Shields, Study Director — Edinburgh Biosciences
Locations (6):
- Romania (6):
  - Institutul Clinic de Urgențe Oftalmologice Prof. Dr. Mircea Olteanu, Bucharest
  - Vedis Ophthalmology Clinic | Ophthalmological Center Dr. Samoila, Cluj-Napoca
  - Dr. Berghian Ophthalmology Clinic, Timișoara
  - Opticlass Clinic, Timișoara
  - Romania Clinica Vista, Ophtalmology Department, Timișoara
  - Spitalul Clinic CF Timisoara, Ophthalmology Department, Timișoara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This is the website of Edinburgh Biosciences, the company sponsoring the clinical studies of the Revisyon medical device. — https://edinburghbiosciences.com/